CLINICAL TRIAL: NCT01951196
Title: Nocturnal Blood Pressure in Chronic Kidney Disease, Obstructive Sleep Apnea and Healthy Subjects - Central and Peripheral 24-h Blood Pressure.
Brief Title: Nocturnal Blood Pressure - Central and Peripheral 24-h Blood Pressure in Chronic Kidney Disease.
Acronym: NOSA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, professor, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Other Study IDs: BGH-1-2013; M-2013-224-13 (Other: The Regional Committee of Health Research Ethics)
Record Dates: First submitted 2013-09-23; First posted 2013-09-26 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Kidney Disease; Obstructive Sleep Apnea
Keywords: Chronic kidney disease; 24 hour blood pressure; central blood pressure; peripheral blood pressure; obstructive sleep apnea
MeSH Terms: conditions — Renal Insufficiency, Chronic; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood, serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic kidney disease, CKD III+IV: 150 patients with Chronic kidney disease, CKD stage III+IV.
- Healthy subjects: 75 healthy subjects.

SUMMARY:
A new study have shown that high nighttime blood pressure (BP) and/or non-dipping (lack of fall in blood pressure during nighttime) is a strong predictor for the risk of cardiovascular disease and mortality in patients with hypertension. Three factors seem to affect the night time blood pressure: chronic kidney disease, obstructive sleep apnea (OSA) or the way ambulatory blood pressure is monitored.

The aim of this study is to analyse the importance of these three factors on nighttime bloodpressure.

Hypothesis:

Central 24 hour blood pressure monitoring provides another measure of daily fluctuations in blood pressure than peripheral 24 hour blood pressure monitoring, because measurement is painless and does not interfere with activities during the daytime or night-time sleep

In chronic kidney disease and OSA the decrease in nocturnal BP is lower than in healthy subjects.

In chronic kidney disease the decrease in the nocturnal BP is inversely correlated to the severity of OSA, the severity of kidney disease, and blood pressure during daytime.

DETAILED DESCRIPTION:
150 patients with chronic kidney disease (CKD III-IV) and 75 healthy subject is examined with both central and peripheral 24 hours blood pressure monitoring, 1 night home polygraphy to determine whether the subject has obstructive sleep apnea, and if so the degree (AHI), blood- and urine samples to determine levels of u-AQP2 og u-ENaCɣ, PRC, p-AngII, p-Aldosterone, p-Avp og p-Endothelin.

ELIGIBILITY:
Patients, group 1:

Inclusion Criteria:

* eGFR 15-59 mL/min/1.73 m2 (estimated GFR)
* 18-80 years
* males and females

Exclusion Criteria:

* lack of desire to participate
* treatment for OSA
* malignant disease
* Abuse of drugs or alcohol
* pregnant and lactating
* incompensated heart failure
* atrial fibrillation
* liver disease (ALAT> 200)
* Severe chronic obstructive lung disease (forced expiratory volume in 1 second <50% predicted)

Healthy Subjects:

inclusion criteria

* Healthy volunteers men and women
* age 40 - 80 years
* BMI within the normal range, ie. between 18.5 to 25.0 kg/m2

exclusion Criteria

* Arterial hypertension, ie. ambulatory blood pressure> 130 mmHg systolic and / or 80 mmHg diastolic.
* a history or clinical signs of cardial, pulmonary, hepato, renal, endocrine, cerebral or neoplastic disorders
* Alcohol abuse, ie. > 14 drinks / week for women and> 21/uge for men
* Substance abuse
* Daily medicine intake/ treatment apart from oral contraceptives
* Smoking
* Pregnancy or breastfeeding
* Lack of desire to participate
* Clinically significant, discrepant results of blood or urine sample at inclusion study (ie B-hemoglobin and B-White blood cell count, p-Sodium, p-Potassium, p-creatinine, p-ALAT, p-bilirubin , p-alkaline phosphatase, p-cholesterol, p-albumin or b-glucose and urine for hematuria, albuminuria or glucosuria)
* Clinically significant differences in the electrocardiogram
* Blood Donation for the past month preceding the day on the first attempt sequence.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Patients with chronic kidney disease, CKD stage III-IV. The patients is followed for their kidney disease at Holstebro Regional Hospital, Denmark, Medical clinic, and the are chosen to participate in the study because of this relation.
  Group 2: Healthy subjects. They arerecruited through postings on public and private companies as well as advertising in local medier.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-12 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
decrease in peripheral systolic blood pressure at night | < 24 hours
  The difference in the decrease in systolic blood pressure at night by peripheral 24-h BP between patients with chronic kidney disease and healthy subjects.

SECONDARY OUTCOMES:
decrease in central systolic blood pressure at night | < 24 hours
  The difference in the decrease in systolic BP at night by central 24-h BP between patients with chronic kidney disease and healthy subjects.
difference in peripheral and central systolic and diastolic blood pressure throughout the day, during the daytime and during nighttime | < 24 hours
  The difference in systolic blood pressure and diastolic blood pressure throughout the day, during the daytime and during nighttime between measurements with peripheral 24-hour monitoring and central 24 hour monitoring in both patients with chronic kidney disease and healthy subjects.
The correlation between the decrease in nighttime blood pressure on the one hand and severity of OSA, severity of kidney disease and blood pressure during the daytime on the other. | < 24 hours
U-AQP2 (urine aquaporin 2) og u-ENaCɣ (urine epithelial sodium channel) | 24 hours
  24 hour urine sample.
PRC (plasma renin concentration), p-AngII (angiotensin II), p-Aldosterone. P-Avp (vasopressin), p-Endothelin. | < 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Research and Medicine, Holstebro Regional Hospital, Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Hornstrup BG, Gjoerup PH, Wessels J, Lauridsen TG, Pedersen EB, Bech JN. Nocturnal blood pressure decrease in patients with chronic kidney disease and in healthy controls - significance of obstructive sleep apnea and renal function. Int J Nephrol Renovasc Dis. 2018 Nov 8;11:279-290. doi: 10.2147/IJNRD.S176606. eCollection 2018. PMID 30510439